CLINICAL TRIAL: NCT04404881
Title: A Phase 2 Study of Bevacizumab for Chronic Bleeding and Iron Deficiency Anemia in Hereditary Hemorrhagic Telangiectasia (Trial Using Systemic Bevacizumab to Treat HHT, TrUST-HHT)
Brief Title: Bevacizumab In Hereditary Hemorrhagic Telangiectasia
Acronym: TrUST-HHT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hanny Al-Samkari, MD (Other)
Responsible Party: Sponsor-Investigator, Hanny Al-Samkari, MD, Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-833
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
Keywords: Hereditary Hemorrhagic Telangiectasia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bevacizumab (Experimental): * The research study procedures include: screening for eligibility, pretreatment period, study treatment, end-of-study visit, and follow-up visit. Each period consists of 12 weeks, for a total of 36 weeks.
  * Pretreatment Period:Hematologic Support: iron transfusions and red cell transfusions as determined by study doctor.
  * Induction Period (first 3 months of bevacizumab treatment):
    * Hematologic Support: iron transfusions and red cell transfusions as determined by study doctor.
    * Bevacizumab: once every 2 weeks via intravenous infusion for up to 12 weeks.
  * Maintenance Period (second 3 months of bevacizumab treatment):
    * Hematologic Support: Iron transfusions and red cell transfusions as determined by study doctor.
    * Bevacizumab: once every 4 weeks via intravenous infusion for up to 12 weeks.
  Interventions: Drug: Bevacizumab (Avastin®)

INTERVENTIONS:
Drug: Bevacizumab (Avastin®) — * Induction Period (first 3 months of bevacizumab treatment):
    -- Bevacizumab: once every 2 weeks via intravenous infusion for up to 12 weeks.
  * Maintenance Period (second 3 months of bevacizumab treatment):
    * Bevacizumab: once every 4 weeks via intravenous infusion for up to 12 weeks.
  Other Names: Avastin®

SUMMARY:
This research study is studying to see whether bevacizumab may treat chronic bleeding and iron deficiency anemia in Hereditary Hemorrhagic Telangiectasia (HHT).

Hereditary Hemorrhagic Telangiectasia (HHT) is a disorder that causes abnormal blood vessel formation. In HHT, there is a mutation in the TGF-β pathway, which results in an increase of vascular endothelial growth factor (VEGF) levels. An increase in VEGF levels can result in poorly formed blood vessels that have a higher rate of bleeding than normal blood vessels. Bevacizumab is designed to block VEGF activity. It is believed that targeting increased VEGF levels may be able to treat HHT.

This research study involves the following study drug:

- Bevacizumab

DETAILED DESCRIPTION:
In this research study, the investigators are studying the study drug, bevacizumab. Researchers would like to see whether bevacizumab effectively treats Hereditary Hemorrhagic Telangiectasia (HHT) and what side effects occur.

- The research study procedures include: screening for eligibility, pretreatment period, study treatment, end-of-study visit, and follow-up visit.

* Participants will be observed for 12 weeks and then receive study treatment for 24 weeks and will be followed for 30 days after ending study treatment.
* This research study involves the following study drug: Bevacizumab
* It is expected that about 33 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating Hereditary Hemorrhagic Telangiectasia (HHT). "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved bevacizumab for Hereditary Hemorrhagic Telangiectasia (HHT), but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria

* A clinical diagnosis of "possible/suspected" or "definite" hereditary hemorrhagic telangiectasia, as defined by presence of 2 or more of the Curacao criteria (spontaneous and recurrent epistaxis, telangiectasias at characteristic sites, visceral arteriovenous malformations (AVMs), first degree relative with HHT).
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of bevacizumab for HHT in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Red blood cell transfusion and/or iron infusion dependence, as defined by a hematologic support score (HSS) of ≥3 in the 3 months prior to consent. HSS is calculated by dividing the total milligrams of elemental iron infused by 250 and adding to this the number of red cell units transfused.
* ECOG performance status ≤2 (see Appendix B).
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes ≥2,000/mcL
  * absolute neutrophil count ≥1,000/mcL
  * platelets ≥50,000/mcL
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN*
  * creatinine ≤ 2.5 mg/dL OR
  * glomerular filtration rate (GFR) ≥45 mL/min/1.73 m2 *Except AST and/or ALT elevation related to HHT-associated hemolytic anemia or liver AVMs, in the opinion of the investigator. Bilirubin thresholds are not included as mild chronic hyperbilirubinemia is common in HHT, likely related to subclinical hemolysis in AVMs. Patients with clinically advanced liver disease should be excluded from participation.
* The effects of bevacizumab on the developing human fetus are unknown. For this reason and because anti-angiogenic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Women should additionally use adequate contraception for the 6 months after discontinuation of bevacizumab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of bevacizumab administration.
* Ability to understand and the willingness to sign a written informed consent document
* Exclusion Criteria
* Participants who have received intranasal or systemic bevacizumab, systemic ramucirumab, or systemic ziv-aflibercept in the 6 weeks prior to consent.
* Participants who have received oral anti-angiogenic agents, including pazopanib, axitinib, sorafenib, thalidomide, lenalidomide, or pomalidomide in the 6 weeks prior to consent.
* Participants receiving oral tranexamic acid or epsilon-aminocaproic acid unless they are on a stable dose for at least 2 weeks prior to consent to be continued at that same dose over the entire duration of the study.
* Participants receiving erythropoiesis-stimulating agents unless they are on a stable dose for at least 4 weeks prior to consent to be continued at that same dose over the entire duration of the study.
* Participants receiving oral iron preparations must discontinue these preparations prior to the initiation of the study (Day 1). Multivitamins or other pharmaceuticals containing iron are allowed if the daily dose of elemental iron does not exceed 25 mg per day.
* Participants receiving systemic estrogen or testosterone preparations unless they are on a stable dose for at least 4 weeks prior to consent to be continued over the entire duration of the study. Use of non-prescription testosterone preparations (e.g. illicit anabolic steroids) in the 4 weeks prior to consent is exclusionary.
* Participants who are receiving any other investigational agents.
* History of allergic reactions to bevacizumab.
* Participants with uncontrolled intercurrent illness, in the opinion of the investigator.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements, in the opinion of the investigator.
* Pregnant women are excluded from this study because bevacizumab is an anti-angiogenic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with bevacizumab, breastfeeding should be discontinued if the mother is treated with bevacizumab. Pregnancy status will be assessed with a serum B-HCG pregnancy test. Women who are menopausal or perimenopausal will have follicle-stimulating hormone levels drawn to confirm menopausal status.
* Known diagnosis of a hypoproliferative anemia (e.g. myelodysplastic syndrome). Nonimmune hemolytic anemia associated with HHT is not exclusionary.
* Significant proteinuria, as defined by a urine protein of >2.0 grams per day (on 24-hour urine protein collection or spot urine protein:creatinine ratio). 24-hour urine protein collection or spot urine protein:creatinine ratio is necessary during screening to quantify urine protein only in patients with screening urine dipstick/urinalysis demonstrates 3+ protein or higher.
* Poorly-controlled hypertension, as defined by a systolic blood pressure >160 mm Hg or diastolic blood pressure >100 mm Hg refractory to medical management.
* Serious or non-healing wound, ulcer or bone fracture.
* Recent hemoptysis, defined as hemoptysis of greater than or equal to one-half teaspoon of blood in the month prior to enrollment.
* Unwillingness to receive red blood cell transfusions and/or intravenous iron infusions according to the hematologic support protocol (HSP) while on study.
* Participants who have surgery planned within 6 months of trial enrollment, or those who have undergone surgery within 1 month of trial enrollment.
* Participants who have received therapeutic endoscopy for gastrointestinal bleeding or nasal surgery for epistaxis within 1 month of trial enrollment.
* Participants who have a history of major thrombophilia, including multiple prior venous and/or arterial thromboembolic events, that in the opinion of the investigator would put them at excessive thrombotic risk.
* Any other medical condition or factor that, in the opinion of the investigator, is likely to interfere with completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in hematologic support score from pretreatment to maintenance | 36 Weeks
  The change in Hematologic Support Score (HSS) from pretreatment to maintenance will be evaluated with a paired t-test or a Wilcoxon signed-rank test, whichever is most appropriate for the distribution of the data. Presence of a statistically-significant difference (P<0.05) will determine if the study achieves its primary outcome measure.

SECONDARY OUTCOMES:
Difference in the individual patient mean hemoglobin | 36 Weeks
  Hemoglobin concentration (g/dL) is the primary clinical measure of red cell mass and blood oxygen-carrying capacity. Hemoglobin thresholds will dictate transfusion on study according to the HSP. Following study completion, for each participant, hemoglobin measurements drawn on day 1 and weeks 2, 4, 6, 8, 10, and 12 will be averaged together to form an average pretreatment hemoglobin and hemoglobin measurements drawn on weeks 24, 26, 28, 30, 32, 34, and 36 will be averaged together to form an average maintenance hemoglobin. Individual patient average pretreatment hemoglobin will be compared to individual patient average maintenance hemoglobin with a paired means comparison test, either a paired ttest or a Wilcoxon signed-rank test, whichever is most appropriate for the distribution of the data.
Difference in the individual patient pRBC transfusion requirement | 36 Weeks
  Number of red cell units transfused will be analyzed separately from iron infusions as a secondary endpoint. The change in number of units of red cells transfused from pretreatment to maintenance will be evaluated with a paired t-test or a Wilcoxon signed-rank test, whichever is most appropriate for the distribution of the data
Difference in the individual patient intravenous iron infusion requirement | 36 Weeks
  Total milligrams of elemental iron infused will be analyzed separately from red cell transfusions as a secondary endpoint. The change in total milligrams of elemental iron infused from pretreatment to maintenance will be evaluated with a paired t-test or a Wilcoxon signed-rank test, whichever is most appropriate for the distribution of the data
Average Maintenance Epistaxis Severity Score | 36 Weeks
  The epistaxis severity score (ESS, not to be confused with the hematologic support score or HSS) is a well-validated, longitudinal, 6-question, 10- point score used specifically to evaluate epistaxis severity in HHT. Individual patient average pretreatment ESS will be compared to individual patient average maintenance ESS with a paired means comparison test, either a paired t-test or a Wilcoxon signed-rank test, whichever is most appropriate for the distribution of the data.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0. | All patients will be evaluable for toxicity from the time of their first treatment with bevacizumab up to 36 weeks
  Number of subjects experiencing grade 3 or higher adverse events (as defined by CTCAE v. 50) and adverse events requiring bevacizumab discontinuation

OTHER OUTCOMES:
HHT-specific Quality of Life Score (HHT-QoL) (exploratory) | 36 Weeks
  Numeric score results of the 4-question HHT-QOL tool from day 1 and week 12 will be averaged together to form an average pretreatment HHT-QOL score and HHT-QOL measurements on weeks 24 and 36 will be averaged together to form an average maintenance HHT-QOL score. The change in HHT-QOL score from pretreatment to maintenance will be evaluated with a paired t-test or a Wilcoxon signed-rank test, whichever is most appropriate for the distribution of the data.
PROMIS Instruments (exploratory) | 36 Weeks
  Three PROMIS instruments [Satisfaction with participation in social roles item bank V1.0 (PROMIS A), Satisfaction with participation in discretionary social activities item bank V1.0 (PROMIS B), and Emotional distress - Depression item bank V1.0 (PROMIS C)] will be administered on day 1, week 12, week 24, and week 36. These PROMIS instruments are chosen given their relevance to HHT symptoms, use in prior HHT QOL study, and high degree of correlation (r=0.6-0.7) with the HHT-QOL instrument being used in this study as well. For each PROMIS instrument, numeric score results of the instrument from day 1 and week 12 will be averaged together to form an average pretreatment score and numeric score results on weeks 24 and 36 will be averaged together to form an average maintenance score. The change in quality of life score from pretreatment to maintenance will be evaluated with a paired t-test or a Wilcoxon signed-rank test, whichever is most appropriate for the distribution of the data.
Hematologic Impact Score (HIS) (exploratory) | 36 Weeks
  Like the HSS, the HIS measures red-cell unit equivalents (RUEs).
  HIS = (Hemoglobin at T2 - HSS at T2) - (Hemoglobin at T1 - HSS at T1)
  For each patient, the HIS will be calculated as follows:
  Hemoglobin at Time 1 (T1) is the hemoglobin at the end of the pretreatment period (week 12 hemoglobin), and hemoglobin at Time 2 (T2) is the hemoglobin at the end of the maintenance period (week 36). The HSS at Time 1 (T1) is the 3-month HSS during the pretreatment period (12 weeks; all hematologic support administered from the day 1 visit [including the date of the day 1 visit] through the week 12 visit [not including support administered on the date of the week 12 visit]) and the HSS at Time 2 (T2) is the 3-month HSS during the maintenance period (12 weeks; all hematologic support administered from the week 24 visit [including the date of the week 24 visit] through the week 36 visit [not including support administered on the date of the week 36 visit]).

CONTACTS AND LOCATIONS:
Overall Officials: Hanny Al-Samkari, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation